CLINICAL TRIAL: NCT01183039
Title: Cellular Effects of Training in Healthy Sedentary Subjects
Brief Title: Effects of Training in Healthy Sedentary Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 5 Santé (Other)
Collaborators: Centre Hospitalier Régional Universitaire Montpellier (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2008-A00209-46
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Sedentary Subjects
Keywords: Sedentary
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventilatory threshold (Active Comparator): Training at the ventilatory threshold
  Interventions: Other: Training
- Metabolic threshold (Active Comparator): Training at the metabolic threshold
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — 20 sessions of training
  Other Names: Vt; Mt

SUMMARY:
The purpose of this study is to understand underlying mechanisms of improved exercise tolerance in Healthy Sedentary Subjects after training program.

DETAILED DESCRIPTION:
Training protocol used is based on recommendations. A minimum of 20 sessions in 4-6 weeks were proposed. The exercise intensity of exercise corresponds to target heart rate at ventilatory threshold measured during incremental exercise test. Training at this intensity allowed us to individualize effort for each patient.

ELIGIBILITY:
Inclusion Criteria:

* healthy Sedentary Subjects

Exclusion Criteria:

* neuromuscular disease
* chronic heart failure
* diabetes
* renal diseases
* liver diseases

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effects of training program on mitochondrial function and oxidative stress | 6 to 8 weeks

SECONDARY OUTCOMES:
Relationship between mitochondrial function, oxidative stress and exercise tolerance in COPD patients | 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maurice MH Hayot, MCU-PH, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (3):
- France (3):
  - Clinique du souffle La valonie, Lodève
  - hopital Arnaud de Vilneuve, Montpellier
  - Clinique du souffle La solane, Osséja